CLINICAL TRIAL: NCT00861991
Title: Enhancing Empathy in Medical Communication Through Perspective-Taking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Benjamin Blatt, GW University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PT2009
Record Dates: First submitted 2009-02-27; First posted 2009-03-16 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Patient Satisfaction
Keywords: medical communication; empathy; medical education; standardized patients; enhancing "patient" satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perspective taking intervention (Experimental): Students were given an instruction to take the perspectives of their standardized patients
  Interventions: Behavioral: Perspective taking instruction
- Control (Active Comparator): Students given standard instructions
  Interventions: Behavioral: Perspective taking instruction

INTERVENTIONS:
Behavioral: Perspective taking instruction — Students were asked to take the perspective of their standardized patients during clinical skills examinations

SUMMARY:
Background: Empathy is critical to clinician-patient communication and patient outcomes. Perspective-taking, an intervention demonstrated in other contexts to induce empathy, has never been studied in a medical context. As a first step in evaluating its potential clinical value, the studies described below assess perspective taking in a series of clinical skills examinations. These examinations are simulated clinical encounters: students encounter and are evaluated by standardized patients (SPs)--actors trained to take on patient roles. Though not real clinical encounters, clinical skills examinations have been demonstrated to test clinical competency well enough to be incorporated into the licensure examination of the National Board of Medical Examiners.

Objective: To assess if perspective-taking improves the satisfaction of standardized patients in three clinical skills examinations.

Hypothesis: Students receiving a perspective taking intervention will receive better standardized patient satisfaction scores than control students.

Design and Setting: Three randomized, controlled studies. Studies 1 and 3: Junior medical students(N = 503), 6-station clinical skills examination. Study 2: physician assistant students (N = 105), 3-station clinical skills examination.

Intervention: The intervention students received a perspective-taking instruction prior to their examination asking them to put themselves in their "patients" shoes and to imagine what they were thinking and feeling. The control students received standard pre-examination instructions. Simulated patients were blind to study condition. Main Outcome Measure: Simulated patient satisfaction scores.

DETAILED DESCRIPTION:
These studies assess the interaction of students and simulated patients (actors)--no real patients were involved.

ELIGIBILITY:
Inclusion Criteria:

* All third year medical and first and second year physician assistant students, George Washington University School of Medicine and Health Sciences

Exclusion Criteria:

* None

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 608 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
standardized patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin C Blatt, MD, Study Director — George Washington University
Locations (1):
- George Washington University School of Medicine, Washington D.C., District of Columbia, United States